CLINICAL TRIAL: NCT00798447
Title: A Prospective, Randomized, Double Blind Study to Compare the Efficacy and Safety of a n-3 Fatty Acid-containing Lipid Emulsion During Parenteral Nutrition in Patients Considered for Major Surgery for Gastric and Colorectal Cancer.
Brief Title: Efficacy and Safety of a PN Regimen Containing n-3 Fatty Acid in Patients Considered After GI Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: B. Braun Melsungen AG (Industry)
Collaborators: B.Braun Taiwan Co., Ltd. (Industry)
Responsible Party: Study Manager, B.Braun Melsungen AG
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HC-G-H-0603
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2011-06

CONDITIONS: GI Cancer
Keywords: post OP
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- lipid emulsion with n-3 FA (Experimental)
  Interventions: Drug: MLF 541
- lipid emulsion without n-3 FA (Active Comparator)
  Interventions: Drug: Lipofundin MCT

INTERVENTIONS:
Drug: MLF 541 — 22-24 h i.v. infusion, maximum 0.75 ml lipid emulsion per kg BW per hour
  Arms: lipid emulsion with n-3 FA
Drug: Lipofundin MCT — 22-24 h iv.infusion, maximum 0.75 ml lipid emulsion per kg BW per hour
  Arms: lipid emulsion without n-3 FA

SUMMARY:
Evaluation of the impact of peri- and post-operative parenteral nutrition enriched with n-3 PUFA on post-operative inflammatory processes.

ELIGIBILITY:
Inclusion Criteria:

* Patients considered for major surgery for gastric and colorectal cancer
* expected requirement for post operative PN or TPN of at least 7 days
* possibility of PN/TPN provision 1 day prior to surgery
* Age >18 years old and <80 years old
* Hemodynamically stable
* Written Informed consent

Exclusion Criteria:

* Participation in a clinical study with an investigational drug or an investigational medical device within one month prior to the start of study
* Patients with sepsis, severe sepsis or septic shock
* Known or suspected drug abuse
* Intrahepatic cholestasis
* General contraindications for infusion therapy such as acute pulmonary edema, hyperhydration and decompensated cardiac insufficiency
* Pregnancy (positive in urine) or lactation
* Autoimmune disease e.g. HIV
* Known hypersensitivity to egg-, soy-, and fish proteins or any of the ingredients of the investigational products
* Hemodynamic failure of any origin (hemorrhagic shock, myocardial infarction, cardiac failure)
* Alterations of coagulation (thrombocytes <150000 /mm3), PT < 50%, PTT > 40 sec
* Ketoacidosis caused by Diabetes mellitus within 7 days prior to onset of study
* Renal insufficiency with serum creatinine > 1.4 mg/dL (>124 µmol/L)
* Patients with severe liver dysfunction with bilirubin >2.5 mg/dL (> 43 µmol/L)
* Lipid disorders, in particular fasting serum triglycerides > 250 mg/dL (>2.85 mmol/L),

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-11; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
reduction of pro inflammatory activity | 30 days

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - National Taiwan University Hospital Taipei, Taipei

REFERENCES:
- [Derived] Ma CJ, Wu JM, Tsai HL, Huang CW, Lu CY, Sun LC, Shih YL, Chen CW, Chuang JF, Wu MH, Wang MY, Lin MT, Wang JY. Prospective double-blind randomized study on the efficacy and safety of an n-3 fatty acid enriched intravenous fat emulsion in postsurgical gastric and colorectal cancer patients. Nutr J. 2015 Jan 21;14:9. doi: 10.1186/1475-2891-14-9. PMID 25609264